CLINICAL TRIAL: NCT01773031
Title: Pancreatic Duct Evaluation in Autoimmune Pancreatitis: Intraindividual Comparison of MR Pancreatography at 3.0 T and 1.5 T
Brief Title: Pancreatic Duct Evaluation in Autoimmune Pancreatitis: MR Pancreatography
Status: Completed | Type: Observational
Sponsor: Jae Ho Byun (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Sponsor-Investigator, Jae Ho Byun, Associate Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMC-2012-1756
Record Dates: First submitted 2013-01-15; First posted 2013-01-23 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Pancreatitis, Chronic; Autoimmune Disease
Keywords: Autoimmune pancreatitis; MR pancreatography
MeSH Terms: conditions — Pancreatitis, Chronic; Autoimmune Diseases; Autoimmune Pancreatitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Autoimmune pancreatitis: Patients with autoimmune pancreatitis based on clinical and CT findings

SUMMARY:
A prospective intra-individual study to compare the image quality of magnetic resonance (MR) pancreatography at 3.0 T and 1.5 T in patients with autoimmune pancreatitis.

DETAILED DESCRIPTION:
Autoimmune pancreatitis (AIP) is a unique form of chronic pancreatitis caused by an autoimmune mechanism that responds well to steroid therapy. One of the most important issues on AIP is to distinguish it from pancreatic cancer as the treatments are totally different from each other. An accurate differentiation of AIP from pancreatic cancer is therefore crucial.

Two most important image findings of AIP are pancreatic enlargement and pancreatic ductal stricture. When CT shows typical diffuse sausage-like swelling of the pancreas and peripancreatic hypodense rim, it is easy to differentiate AIP from pancreatic cancer. However, those typical cases are not very common and, moreover, 30% of AIP manifest as focal mass/enlargement of the pancreas, making a differential diagnosis very difficult. When pancreatic feature is atypical at CT, it is important to find diffuse or multifocal stricture of the main pancreatic duct that is characteristic feature of AIP. In AIP, a diffusely attenuated pancreatic duct is thinner than normal, and this does not appear at CT. Pancreatography is therefore necessary.

Two current imaging tools to demonstrate the pancreatic duct are endoscopic retrograde pancreatography (ERP) and MR pancreatography (MRP). ERP provides high resolution images using different projections and enables various procedures including aspiration/biopsy and stent insertion. However, the use of diagnostic ERP in diagnosing AIP has been debated as ERP is an invasive procedure, having potential complications including pancreatitis, perforation of the stomach or duodenum. Moreover, it is difficult to perform endoscopic procedure in patients who underwent gastric surgery. Whereas, MRP can noninvasively image the pancreatic and biliary systems at the same time without risks of procedure-related complications and can evaluate other intrabdominal organs on cross-sectional images. The relatively lower spatial resolution of MRP using 1.5 T compared with ERP images may make it difficult to demonstrate fine changes of the pancreatic duct in AIP and sometimes make false positive or negative findings.

The superiority of 3.0 T over 1.5 T MR systems has been observed in several studies. However, only a few studies using the 3.0 T MR systems in the pancreaticobiliary tract have been reported and, furthermore, the usefulness of 3.0 T MRP for the diagnosis of AIP has not yet been investigated.

The purpose of this study is to prospectively compare the image quality of MRP at 3.0 T and 1.5 T in patients with AIP using ERP as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Typical CT findings (diffuse sausage-like pancreatic swelling or multifocal pancreatic swelling with or without peripancreatic rim, multifocal biliary stricture, renal lesion, or retroperitoneal fibrosis)
* Serum level of immunoglobulin G fraction 4 > 135mg/dL

Exclusion Criteria:

* Patients under 20 years of age
* Women who are pregnant, lactating or who are of childbearing potential
* Patients with any physical or mental status that interferes with the signing of informed consent
* Patients with a contraindication for MRP or ERP examination

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with probable autoimmune pancreatitis based on clinical and CT findings
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Scoring for visualization of the main pancreatic duct on 1.5 T and 3.0 T MRP | Outcome measure will be assessed after a week following MRP examination
  1. Scoring for overall visualization of the main pancreatic duct (MPD): 1-4 points (1, entirely invisible; 2, faintly and partially visible; 3, faintly but entirely visible/clearly but partially visible; 4, clearly and entirely visible)
  2. Scoring for visualization of MPD stricture: 1-4 points (1, invisible; 2, poorly visible; 3, moderately visible; 4, clearly visible)
     * Reference standard: ERP

SECONDARY OUTCOMES:
Signal-to-noise ratio of the main pancreatic duct on 1.5 T and 3.0 T MRP | Outcome measure will be assessed after a week following MRP examination
The rate of concordance in the stricture type of the main pancreatic duct between MRP and ERP | Outcome measure will be assessed after a week following MRP examination
  Stricture type of the main pancreatic duct: 1, diffuse; 2, segmental; 3, focal; 4, multifocal
Scoring for confidence in diagnosing AIP based on MRP findings | Outcome measure will be assessed after a week following MRP examination
  Scoring for confidence: 1-4 points (1, low probability; 2, indeterminate probability; 3, moderate probability; 4, high probability)

CONTACTS AND LOCATIONS:
Overall Officials: Jae Ho Byun, MD, PhD, Principal Investigator — University of Ulsan College of Medicine, Asan Medical Center
Locations (1):
- Division of Abdomen, Department of Radiology & Research Institute of Radiology, University of Ulsan College of Medicine, Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Finkelberg DL, Sahani D, Deshpande V, Brugge WR. Autoimmune pancreatitis. N Engl J Med. 2006 Dec 21;355(25):2670-6. doi: 10.1056/NEJMra061200. No abstract available. PMID 17182992
- [Background] Kim JH, Kim MH, Byun JH, Lee SS, Lee SJ, Park SH, Lee SK, Park DH, Lee MG, Moon SH. Diagnostic Strategy for Differentiating Autoimmune Pancreatitis From Pancreatic Cancer: Is an Endoscopic Retrograde Pancreatography Essential? Pancreas. 2012 May;41(4):639-647. doi: 10.1097/MPA.0b013e31823a509b. Epub 2012 Jan 5. PMID 22228050
- [Background] Park SH, Kim MH, Kim SY, Kim HJ, Moon SH, Lee SS, Byun JH, Lee SK, Seo DW, Lee MG. Magnetic resonance cholangiopancreatography for the diagnostic evaluation of autoimmune pancreatitis. Pancreas. 2010 Nov;39(8):1191-8. doi: 10.1097/MPA.0b013e3181dbf469. PMID 20467343
- [Background] Onishi H, Kim T, Hori M, Murakami T, Tatsumi M, Nakaya Y, Nakamoto A, Osuga K, Tomoda K, Nakamura H. MR cholangiopancreatography at 3.0 T: intraindividual comparative study with MR cholangiopancreatography at 1.5 T for clinical patients. Invest Radiol. 2009 Sep;44(9):559-65. doi: 10.1097/RLI.0b013e3181b4c0ae. PMID 19692840